CLINICAL TRIAL: NCT06828913
Title: Effect of Social Media on Parental Oral Health Promotion ; a Pre and Post Test Design
Brief Title: Effect of Social Media on Parental Oral Health Promotion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Sayed Ahmed, the principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: social media in oral health
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: The Study Focus on the Role of Social Media on Promoting Parental Oral Health
Keywords: social media , parental oral health; social media; pre and post study desgin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A group of parent of children (Other): a group of parent of children on online platforms
  Interventions: Other: Oral Health information on online platforms

INTERVENTIONS:
Other: Oral Health information on online platforms — oral health

SUMMARY:
The study aims to measure the effectiveness of social media in raising parental oral health awareness.

DETAILED DESCRIPTION:
Health Education is a key element in Health promotion. Oral health awareness has a pivotal role in community prevention programs. The methods used for health education have developed through the years to fit the population's needs and to cope with the technological revolution. Nowadays social media has become the easiest, fastest, and most acceptable portal for people. However the benefits of social media are huge for health communication, the shared information should be assessed and monitored for quality and reliability and the privacy of the users should be secured, up to our knowledge there is no reliable source for education on promoting oral health on the social media platform in our community, Although the traditional methods to educate parent like visiting the dentist are more common, Studies show that parents and children had little recollection of any preventive oral health conversations when visiting the dentist. we use oral health Information based on AAPD guidelines that we be provided on social media platforms and then measure the effectiveness of social media in raising parental oral awareness

ELIGIBILITY:
Inclusion Criteria:

1. Parents who volunteer to participate
2. parent have access to social media networks & smartphone.
3. Parents of infants and toddlers
4. parents of primary school children.

Exclusion Criteria:

1. parent who do not volunteer to participate
2. parent have Low educational standard (unable to use smartphones).
3. Parent of middle school children

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Parental oral health Knowledge, attitude, and practice | 2 month
  we will measure the parental oral health knowledge , attitude and practice the measuring device online questionnaire measuring unit percentage from (0 - 100 )

SECONDARY OUTCOMES:
parental Satisfaction | 2 month
  we will measure the parental satisfaction measuring device : online questionnaire only after study completed measuring unit percentage (0 -100)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 8- Ganji, K.K., Patil, S., Alhadi, A. and Alhadi, M., 2018. Parent's Knowledge, Attitude and Practice on Prevention of Early Childhood Caries in Al jouf Province, Saudi Arabia. Pesquisa Brasileira em Odontopediatria e Clínica Integrada,
- [Background] Shah AH, Refeai MA, Alolaywi FM, Gulzar S, Asiri FY, Jameel ABA. Satisfaction of Oral Health Education among Parents and Caregivers Regarding Children with Special Healthcare Needs in Riyadh, Saudi Arabia. J Contemp Dent Pract. 2021 Aug 1;22(8):894-899. PMID 34753841
- [Background] 6- Singh, S., Saraf, B.G., Sheoran, N., Singh, R. and Kapil, D., 2023. Knowledge, Attitude, and Practice of Parents about Child's Oral Health in Faridabad and its Correlation with Prevalence of Dental Caries in Children through a Questionnaire Survey. Indian Journal of Dental Sciences, 15(3), pp.151-156.
- [Background] Ahovuo-Saloranta A, Forss H, Walsh T, Hiiri A, Nordblad A, Makela M, Worthington HV. Sealants for preventing dental decay in the permanent teeth. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD001830. doi: 10.1002/14651858.CD001830.pub4. PMID 23543512
- [Background] Sharma S, Mohanty V, Balappanavar AY, Chahar P, Rijhwani K. Role of Digital Media in Promoting Oral Health: A Systematic Review. Cureus. 2022 Sep 7;14(9):e28893. doi: 10.7759/cureus.28893. eCollection 2022 Sep. PMID 36225421